CLINICAL TRIAL: NCT03461731
Title: Investigation of the Role of 905-nm Laser Light in the Delay of Muscle Fatigue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: College of Charleston (Other)
Responsible Party: Principal Investigator, Linda Ramball Jones, Professor of Physics, College of Charleston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: IRB-2017-01-03-123913
Record Dates: First submitted 2018-02-27; First posted 2018-03-12 (Actual); Last update posted 2018-03-12 (Actual); Status verified 2018-03

CONDITIONS: Muscle Fatigue
Keywords: Low-Level Light Therapy
MeSH Terms: interventions — Lasers

STUDY DESIGN:
Intervention Model Description: Each participant receives placebo and two different light treatments in random order
Who Masked: Participant
Masking Description: The participant cannot tell if the laser is turned on because the fan runs for the placebo as well
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (4):
- Control (Sham Comparator): Participant will receive a sham treatment that consists of just the 660-nm aiming beam
  Interventions: Device: Control
- 800 nm laser (Experimental): 800 nm laser will be applied at 4.4 Joules per square cm on the forearm during 40 repetitive hand grips
  Interventions: Device: 800 nm laser
- combination laser (Experimental): 905 nm and 800 nm will be applied at 4.4 joules per square cm with a total of 8.8 Joules per square cm during 40 repetitive handgrips.
  Interventions: Device: combination laser
- 905 nm laser (Experimental): 905 nm laser will be applied at 4.4 Joules per square cm on the forearm during 40 repetitive hand grips
  Interventions: Device: 905 nm laser

INTERVENTIONS:
Device: Control — laser beam only
  Arms: Control
Device: 800 nm laser — 800 nm laser applied to forearm at 4.4 Joules per square cm during 40 hand grips
  Arms: 800 nm laser
Device: combination laser — 800 nm and 905 nm laser applied to forearm at 4.4 Joules per square cm during 40 hand grips
  Arms: combination laser
Device: 905 nm laser — 905 nm laser applied to forearm at 4.4 Joules per square cm during 40 hand grips
  Arms: 905 nm laser

SUMMARY:
800-nm laser light has been shown to delay muscle fatigue when applied before exercise. The effect of illumination during the aerobic phase of strenuous exercise has not been studied. The investigators hypothesize that the increased energy donated to cells during the aerobic phase will significantly delay muscle fatigue. A novel aspect of this study is to include simultaneous treatment with near infrared light at 800 nm and 905 nm. Fatigue index and change in lactate blood level will be used to compare the different laser treatments for each participant. Monte Carlo simulations of light energy reaching the muscle will be carried out, based on skin-fold thickness measurements of each participant. The investigators believe this will be the first report of optical dosimetry as a function of adipose thickness and it will enable estimation how much of the light applied to the skin surface is able to penetrate to the muscles that are thought to be affected. The results of this study will help clinicians to optimize treatment for individual patients.

DETAILED DESCRIPTION:
Rationale, Objectives and Significance A recent study has shown that low intensity Near Infrared (NIR) light at 810 nm applied before exercise results in an increase in performance and decrease in oxidative stress and muscle damage (1). Another study by the same group with 830 nm light showed a delay in exercise-induced muscle fatigue when applied before exercise (2). A number of studies have shown varying results with near infrared light for pain relief, inflammation and wound healing. The results often vary in part due to the difference in the wavelength and intensity of the light source and variation in the depth of penetration of the light. Red and NIR light is known to penetrate significantly into biological tissues. For example, a recent study presents qualitative evidence that 830 nm light penetrated significantly through cadaver soft tissue and a human hand in vivo (3). The optical properties of various human tissues have been studied at 800 to 950 nm so it is possible for the investigators to calculate the precise distribution of near infrared light in relation to the physiological effects. The investigators are well equipped to carry this out with an original, calibrated Monte Carlo program. The mechanism of action for low intensity red to NIR light has been fairly well studied and is thought to occur through absorption of the light by mitochondrial cytochrome c oxidase which leads to energy production in the illuminated cells (4). The effect of illumination DURING the aerobic phase of strenuous exercise has not been studied. The investigators hypothesize that the increased energy donated to cells during the aerobic phase will significantly delay muscle fatigue.

fatigue index and lactate blood level will be used to compare the different laser treatments. Another novel aspect of this study is to include NIR light at 905 nm. A hypothesized mechanism for delay of muscle fatigue is a light-initiated release of oxygen from hemoglobin molecules by 905-nm laser light, resulting in increased oxygenation of the local tissue. The laser may heat the tissue slightly so it is not clear whether oxygen release is due to a thermal or photochemical mechanism. A recent study of low level light (660 nm, 350 mW, 15 minutes) resulted in no measurable change in local tissue oxygenation for healthy participants (5). Another recent study with a more intense light source (K-laser at 800, 907 and 970 nm, 3 W, 4 minutes) demonstrated increased blood flow in the upper arm following irradiation with the NIR laser (6). However the authors did not measure the temperature of the irradiated tissue.

In the proposed study the investigators will keep the intensity of 800 nm light constant in all of the trials. The proposed study will include collection of surface temperature during the treatment to begin to document whether tissue heating is involved in the mechanism. The adipose thickness (calculated from skin fold thickness) will be used with the Monte Carlo simulation to calculate the fraction of light that is expected to reach the muscle for each participant. This will be the first report of optical dosimetry as a function of adipose thickness and it will enable estimation of how much of the light applied to the skin surface is able to penetrate to the muscles that are thought to be affected. The results of this study will help clinicians to optimize treatment for individual patients.

1. Thiago de Marchi, Ernesto Cesar Pinto Leal Junior et al, Low level laser therapy (LLLT) in human progressive intensity running: effects on exercise performance, skeletal muscle status and oxidative stress. (2012) Lasers in Medical Science 27:231236.
2. Ernesto Cesar Pinto Leal Junior, Rodrigo Alvaro Brandao LopexMartins et al. Effect of 830nm lowlevel therapy in exercise induced skeletal muscle fatigue in humans. (2009) Lasers in Medical Science 24:425431.
3. Jared Jagdeo, Lauren Adams, et al. Transcranial red and near infrared light transmission in a cadaveric model. (2012) PLOS ONE 7:10 e47460
4. Janis Eells, Margaret WongRiley, et al. Mitochondrial signal transduction in accelerated wound and retinal healing by near infrared light therapy. (2004) Mitochondrion Sep; 4(56):55967.
5. Franziska Heu, Clemens Forster, Barbara Namer, Adrian Dragu, Werner Lang. Effect of lowlevel laser therapy on blood flow and oxygenhemoglobin saturation of the foot skin in healthy subjects: a pilot study. (2013) Laser Therapy 22(1): 2130.
6. Kelly Larkin, Jeffrey Martin, Elizabeth Zeanah, Jerry Tue, Randy Braith, Paul Borsa. Limb blood flow after class 4 laser therapy. (2012) Journal of Athletic Training. 47(2): 178183.

ELIGIBILITY:
Inclusion Criteria

* Between the ages of 18 and 25 years

Exclusion Criteria

* Upper extremity surgery
* Upper body musculoskeletal injury to the non-dominant arm within the past year
* Tattoos on the forearm
* Photosensitizing medications (listed on the consent form)

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2017-02-20 (Actual); Primary Completion 2017-07-30 (Actual); Study Completion 2017-07-31 (Actual)

PRIMARY OUTCOMES:
Muscle fatigue | Muscle fatigue is calculated from force data immediately after each treatment.
  Grip force measured by a dynamometer

SECONDARY OUTCOMES:
Lactate | Lactate is measured immediately before each laser treatment and three minutes after each treatment.
  Change in blood lactate level

CONTACTS AND LOCATIONS:
Overall Officials: Linda R Jones, Ph.D., Principal Investigator — College of Charleston
Locations (1):
- College of Charleston, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after de-identification
Supporting Information: Study Protocol
Time Frame: immediately following publication. No end date
Access Criteria: Anyone who wishes to access the data

REFERENCES:
- [Background] De Marchi T, Leal Junior EC, Bortoli C, Tomazoni SS, Lopes-Martins RA, Salvador M. Low-level laser therapy (LLLT) in human progressive-intensity running: effects on exercise performance, skeletal muscle status, and oxidative stress. Lasers Med Sci. 2012 Jan;27(1):231-6. doi: 10.1007/s10103-011-0955-5. Epub 2011 Jul 8. PMID 21739259
- [Background] Leal Junior EC, Lopes-Martins RA, Vanin AA, Baroni BM, Grosselli D, De Marchi T, Iversen VV, Bjordal JM. Effect of 830 nm low-level laser therapy in exercise-induced skeletal muscle fatigue in humans. Lasers Med Sci. 2009 May;24(3):425-31. doi: 10.1007/s10103-008-0592-9. Epub 2008 Jul 23. PMID 18649044
- [Background] Jagdeo JR, Adams LE, Brody NI, Siegel DM. Transcranial red and near infrared light transmission in a cadaveric model. PLoS One. 2012;7(10):e47460. doi: 10.1371/journal.pone.0047460. Epub 2012 Oct 15. PMID 23077622
- [Background] Eells JT, Wong-Riley MT, VerHoeve J, Henry M, Buchman EV, Kane MP, Gould LJ, Das R, Jett M, Hodgson BD, Margolis D, Whelan HT. Mitochondrial signal transduction in accelerated wound and retinal healing by near-infrared light therapy. Mitochondrion. 2004 Sep;4(5-6):559-67. doi: 10.1016/j.mito.2004.07.033. PMID 16120414
- [Background] Heu F, Forster C, Namer B, Dragu A, Lang W. Effect of low-level laser therapy on blood flow and oxygen- hemoglobin saturation of the foot skin in healthy subjects: a pilot study. Laser Ther. 2013;22(1):21-30. doi: 10.5978/islsm.13-or-03. PMID 24155546
- [Background] Larkin KA, Martin JS, Zeanah EH, True JM, Braith RW, Borsa PA. Limb blood flow after class 4 laser therapy. J Athl Train. 2012 Mar-Apr;47(2):178-83. doi: 10.4085/1062-6050-47.2.178. PMID 22488283